CLINICAL TRIAL: NCT01847001
Title: A Study of the Beta-blocker Propranolol Alone and With Chemotherapy in Patients Receiving Neoadjuvant Treatment for Newly Diagnosed Breast Cancer
Brief Title: Study of Propranolol in Newly Diagnosed Breast Cancer Patients Undergoing Neoadjuvant Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAI9158; UL1TR000040 (NIH)
Record Dates: First submitted 2013-04-23; First posted 2013-05-06 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Malignant Neoplasm; Breast Cancer
Keywords: Breast Cancer; Neoadjuvant; Experimental; Biomarker; Breast imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Propranolol; propranolol CR; Paclitaxel; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Trastuzumab; pertuzumab; Doxorubicin; Cyclophosphamide; Surgical Procedures, Operative; Premedication; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propranolol + Neoadjuvant Chemotherapy (Experimental): Subjects will receive 2 types of chemotherapy regimens plus propranolol treatment.
  * Regimen I, involves paclitaxel (may be substituted with nab-paclitaxel; maybe given with premedication), and
  * Regimen II involves doxorubicin (maybe given with anti-nausea therapy) and cyclophosphamide (maybe given with Pegfilgrastim).
  * If your tumor is HER2 positive, you will also receive trastuzumab and pertuzumab.
  After you complete all chemotherapy plus propranolol treatment, you will then have surgery to remove the breast tumor.
  DOT imaging will be done at 4 additional time points, including beo.
  Interventions: Drug: Propranolol; Other: DOT imaging; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Procedure: Surgery; Drug: Premedication; Drug: Anti-nausea therapy; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Propranolol — Propranolol starting dose is 20mg b.i.d.; propranolol dose is up-titrated to 40mg b.i.d. to 80 mg daily with chemotherapy depending on tolerability. Tolerability is assessed every 2 weeks.
  Other Names: Inderal; Inderal LA ®; InnoPran XL ®
Other: DOT imaging — (Non-experimental) During the baseline visit, you will undergo DOT evaluation of your tumor for determination of blood, fat, and water content in the affected and unaffected breast. DOT readings will be obtained at 4 additional time points: after paclitaxel week #3, before AC week #1, before AC week #3, and prior to surgery.
  Other Names: Breast imaging - Diffuse Optical Tomography (DOT)
Drug: Paclitaxel — (Non-experimental) given as a one-hour intravenous infusion (IV) every week for a total of 12 weeks; the first dose of paclitaxel may be given over 90 minutes, per the discretion of your treating doctor. The dose will be given in 80 mg/m2 based on individual body surface area (BSA). This drug is given through a vein in the arm or a catheter (eg. Infusaport, Portacath).
  Other Names: Abraxane
Drug: Nab-paclitaxel — (Non-experimental) In the event paclitaxel is not available due to manufacturing and supply shortages, nab-paclitaxel will be substituted for paclitaxel. The dose is 100 mg/m2 IV infusion over 30 minutes weekly (or institutional standard). No premedications are given with nab-paclitaxel.
  Other Names: Abraxane
Drug: Trastuzumab — (Non-experimental) (only if HER2-positive): Trastuzumab is given as an IV infusion initially over 90 minutes for the first dose, then 30-60 minutes every 3 weeks in subsequent doses if well tolerated. To be given every 3 weeks with paclitaxel/propranolol.
  Other Names: Herceptin
Drug: Pertuzumab — (Non-experimental) (only if HER2-positive): Pertuzumab is given as an IV infusion over 60 minutes on the first dose, then 30-60 minutes every 3 weeks if well tolerated. To be given every 3 weeks with paclitaxel/propranolol.
  Other Names: Perjeta
Drug: Doxorubicin — (Non-experimental) Doxorubicin will be given as a 510 minute intravenous infusion (IV) in a dose of 60 mg/m2; cyclophosphamide will be given as a 3060 minutes intravenous infusion (IV) in a dose of 600 mg/m2 based on BSA. This chemotherapy regimen will be given every 2 weeks for total of 8 weeks or 2 months.
  Other Names: Adriamycin
Drug: Cyclophosphamide — (Non-experimental) Doxorubicin 60 mg/m2 IV over 5-10 minutes, Cyclophosphamide 600 mg/m2 IV infusion over 30-60 minutes. The first cycle should be initiated with 3 weeks after the last paclitaxel and/or trastuzumab/pertuzumab dose.
  Other Names: AC
Procedure: Surgery — After you complete all chemotherapy plus propranolol treatment, you will then have surgery to remove the breast tumor if your doctor feels that it is medically appropriate (if you have had a good response to the treatment) - lumpectomy/mastectomy.
  Other Names: No other name
Drug: Premedication — As premedication to prevent some of the side effects associated with paclitaxel, you will also receive dexamethasone (Decadron) in a dose of 10 mg, diphenhydramine (Benadryl) in doses of 2550 mg, and an H2 blocker (eg. ranitidine 50 mg or equivalent) 3060 minutes before each paclitaxel infusion. If no hypersensitivity reactions are experienced, dexamethasone may be reduced in increments of 2 mg per week per dose (until a minimum of 2 mg has been reached).
  Other Names: No other name
Drug: Anti-nausea therapy — In addition to doxorubicin, you will receive an anti-nausea therapy and dexamethasone about 3060 minutes before AC chemotherapy.
  Other Names: No other name
Drug: Pegfilgrastim — When you receive the AC chemotherapy, you will also receive treatment with a drug called pegfilgrastim (Neulasta). Neulasta is a commercially available drug. It stimulates the production of white blood cells and reduces the likelihood of developing a low white blood cell count and fever after chemotherapy. It will be given as an injection under the skin on the day after each chemotherapy treatment (day 2).
  Other Names: Neulasta

SUMMARY:
This study is being conducted in patients with newly diagnosed breast cancer that will be undergoing chemotherapy prior to surgery - neoadjuvant chemotherapy. The study involves treatment with standard chemotherapy and a commonly used, FDA-approved, blood pressure drug called propranolol (Inderal). The purposes of this study are to:

1. Determine the effect of propranolol plus chemotherapy on breast cancer cells as well as the growth of blood vessels surrounding breast cancer cells.
2. Determine the side effect profile of propranolol and chemotherapy in patients with breast cancer receiving neoadjuvant chemotherapy.

This research is being done because previous laboratory work has shown that propranolol may decrease the ability for the blood vessels around breast cancer cells to grow, which may be important in helping cancer cells grow. It also may reduce the likelihood for breast cancer cells to spread. If changes are seen in the breast cancer cells and surrounding blood vessels in this study, we will pan to evaluate whether propranolol decreases the likelihood of breast cancer from recurring in future, later studies. All chemotherapy regimens used in this study have been the standard of care for many years; however, the use of propranolol is being researched along with the chemotherapy regimens.

DETAILED DESCRIPTION:
While a number of therapeutic options exist for patients with breast cancer (BC), breast tumor biology is differs across tumors and not all BCs respond to treatment. Identifying a marker predicting response could spare non-responders unnecessary side effects, cost, and time. A recent example in BC is bevacizumab, an expensive anti-angiogenic monoclonal antibody, for which the FDA revoked approval for patients with metastatic BC. While this targeted therapy may benefit some patients, no appropriate predictive marker has been identified in the drug development process. An ideal biologic marker would be easy to perform, reliable, low-cost and non-invasive. A limitation of assessing tumor-based markers in metastatic BC is the inability to procure tumor tissue at different treatment times. To circumvent this issue, anti-cancer agents can be assessed pre-operatively, where women with newly diagnosed BC receive a study drug, alone or with chemotherapy, between diagnostic breast biopsy and surgical resection. In addition, tumor changes can be directly compared to modulation of non-invasive markers, such as functional radiographs or blood, to identify a non-invasive marker predicting tumor response.

The investigators are conducting a neoadjuvant single-institution trial with the non-selective, inexpensive β -blocker propranolol with chemotherapy in locally advanced BC. β-blockade regulates angiogenesis in primary breast tumors. In these trials, the investigators plan to evaluate treatment-related microvascular response via changes in breast Diffuse Optical Tomography (DOT), a non-invasive, fast, safe, and inexpensive breast imaging tool. As the optical property contrast from endogenous chromophores (oxyhemoglobin, deoxyhemoglobin, water, and lipid) provides information on tissue vascularity, it can monitor response to anti-angiogenic agents. DOT changes occur as early as 1 week after starting pre-operative therapy. The dynamic DOT system incorporated in these trials is unique to Columbia University Medical Center (CUMC), as it has been designed by Columbia biomedical engineers. CUMC's laboratory collaborators have measured this DOT system with anti-angiogenesis agents in animal models, demonstrating the translational nature of this project. While non-dynamic DOT has been assessed in other neoadjuvant trials with small cohorts receiving heterogeneous chemotherapy agents, none have evaluated DOT response to anti-angiogenic agents.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking women age ≥18
* Heart Rate > 60 bpm
* Systolic Blood Pressure > 100 mm/Hg
* Deemed eligible to receive neoadjuvant chemotherapy with 12 cycles of weekly taxane therapy (paclitaxel 80mg/m2 or Abraxane 100 mg/m2 if there is a shortage of paclitaxel) followed by 4 cycles of Adriamycin (60mg/m2) and cyclophosphamide (600 mg/m2) given every 2 weeks with growth-factor support.
* Echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) with ejection fraction > 50%.
* Patients with hormone receptor +/- and human epidermal growth factor receptor 2 protein (HER2) +/- breast cancer are eligible
* If a patient has HER2-positive breast cancer, Herceptin and Perjeta will be given along with taxane therapy
* Any stage invasive breast cancer provided the primary breast tumor size is ≥ 1 cm
* Agree to participate in research blood collection at 4 different time periods (20 ml = 4 teaspoons)
* Agree to the evaluation of already collected core biopsy, as well as surgical resection tissue, for predictive biomarkers. The biopsy prior to Taxol #1 is optional.

Exclusion Criteria:

* Patients failing to meet the inclusion criteria
* Corrected QT interval (QTc) prolongation as defined by > 470 milliseconds on electrocardiogram (ECG)
* First-degree Atrioventricular (AV) block on ECG in which P-R interval lengthened > 200 milliseconds; Second Degree; or Third Degree
* On beta-blocker treatment. If discontinued, patients must have been off beta-blockers for at least 3 months.
* History of asthma, given concern for β-blockade in this population

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2018-12-31 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M. Kalinsky, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Propranolol + Neoadjuvant Chemotherapy: Subjects will receive 2 types of chemotherapy regimens plus propranolol treatment.
  * Regimen I, involves paclitaxel (may be substituted with nab-paclitaxel; maybe given with premedication), and
  * Regimen II involves doxorubicin (maybe given with anti-nausea therapy) and cyclophosphamide (maybe given with Pegfilgrastim).
  * If your tumor is HER2 positive, you will also receive trastuzumab and pertuzumab.
  After you complete all chemotherapy plus propranolol treatment, you will then have surgery to remove the breast tumor.
  DOT imaging will be done at 4 additional time points, including beo.
  Propranolol: Propranolol starting dose is 20mg b.i.d.; propranolol dose is up-titrated to 40mg b.i.d. to 80 mg daily with chemotherapy depending on tolerability. Tolerability is assessed every 2 weeks.
Period: Overall Study
Arm/Group | Propranolol + Neoadjuvant Chemotherapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Propranolol + Neoadjuvant Chemotherapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Systolic Blood Pressure Measured [Mean (Full Range); unit: mmHg] | 121.7 [107 to 138]
Average Heart Rate (HR) [Mean (Full Range); unit: bpm] | 76.8 [61 to 94]

OUTCOME MEASURES:

1. Primary Outcome: Mean Adherence to Propranolol
Description: Propranolol adherence was documented biweekly by pill counts and drug diary checks.
Time Frame: Approximately 6 months
Measure: Mean (Full Range); unit: Percentage of propanolol adherence
Arm/Group | Propranolol + Neoadjuvant Chemotherapy
Number analyzed (Participants) | 10
Percentage of propanolol adherence | 96 [89 to 100]

2. Primary Outcome: Total Number of Participants Who Reached The Target Propranolol Dosing
Description: The target Propranolol dosing was 80mg ER daily.
Time Frame: Approximately 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Propranolol + Neoadjuvant Chemotherapy: Subjects will receive 2 types of chemotherapy regimens plus propranolol treatment.
  * Regimen I, involves paclitaxel (may be substituted with nab-paclitaxel; maybe given with premedication), and
  * Regimen II involves doxorubicin (maybe given with anti-nausea therapy) and cyclophosphamide (maybe given with Pegfilgrastim).
  Propranolol: Propranolol starting dose is 20mg b.i.d.; propranolol dose is up-titrated to 40mg b.i.d. to 80 mg daily with chemotherapy depending on tolerability. Tolerability is assessed every 2 weeks.
Arm/Group | Propranolol + Neoadjuvant Chemotherapy
Number analyzed (Participants) | 10
Participants | 9

3. Secondary Outcome: Number of Patients With Pathologic Complete Response
Description: Response was confirmed with pathology.
Time Frame: Approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol + Neoadjuvant Chemotherapy
Number analyzed (Participants) | 10
Participants | 1

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events will be collected/analyzed and reported by December 2020.
Arm/Group | Propranolol + Neoadjuvant Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol + Neoadjuvant Chemotherapy (N=10)
Colitis (Gastrointestinal disorders) | 1 (1) — Grade 3 requiring hospital admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol + Neoadjuvant Chemotherapy (N=10)
Fatigue (General disorders) | 2 (2) — Grade 2
QTc prolongation (Cardiac disorders) | 2 (2) — Grade 2 but asymptomatic
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Central line infection (Infections and infestations) | 1 (1) — Grade 3
Infusion Reaction (General disorders) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT01847001/Prot_SAP_000.pdf